CLINICAL TRIAL: NCT05384873
Title: Multicentre, Randomised, Open-label, Parallel-group Trial to Evaluate Immunonutrition in Improving Efficacy of Immunotherapy in Patients With Metastatic Non-small Cell Lung Cancer, Undergoing Systematic Nutritional Counseling
Brief Title: Immunonutrition for Improving the Efficacy of Immunotherapy in Patients With Metastatic Non-small Cell Lung Cancer
Acronym: MURAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: San Luigi Gonzaga Hospital (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Riccardo Caccialanza, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0020364/22
Record Dates: First submitted 2022-05-09; First posted 2022-05-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunonutrition (Experimental): In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement enriched in immunonutrients (Oral Impact®). The intervention will start approximately two weeks before anticancer treatment initiation and will continue up to first disease re-assessment (12-14 weeks) and prolonged according to patient's needs
  Interventions: Dietary Supplement: Immunonutrition
- Control dietary intervention (Active Comparator): Patients will receive nutritional counseling as standard of care. Nutritional counseling may comprise the use of oral nutritional supplements (ONS), which are usually prescribed when patients are unable to maintain satisfactory spontaneous food intake (less than 50% of the requirement for more than one week or only 50-75% of the requirement for more than two weeks). Therefore, in this arm the use of isonitrogenous standard blend ONS will be considered according to the regular assessment of food intake.
  Interventions: Other: Control dietary intervention

INTERVENTIONS:
Dietary Supplement: Immunonutrition — In addition to nutritional counseling, patients will receive two servings of an oral high-calorie-high-protein nutritional liquid supplement enriched in immunonutrients (Oral Impact®). The intervention will start approximately two weeks before anticancer treatment initiation and will continue up to first disease re-assessment (12-14 weeks) and prolonged according to patient's needs
  Arms: Immunonutrition
Other: Control dietary intervention — Patients will receive nutritional counseling as standard of care. Nutritional counseling may comprise the use of oral nutritional supplements (ONS), which are usually prescribed when patients are unable to maintain satisfactory spontaneous food intake (less than 50% of the requirement for more than one week or only 50-75% of the requirement for more than two weeks). Therefore, in this arm the use of isonitrogenous standard blend ONS will be considered according to the regular assessment of food intake.
  Arms: Control dietary intervention

SUMMARY:
The present study was designed to evaluate the efficacy of the early systematic provision of oral nutritional supplements enriched in immunonutrients in non-small lung cancer patients undergoing immunotherapy and receiving nutritional counseling

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histological diagnosis of metastatic non-small cell lung cancer (both squamous and non-squamous histology);
* First-line treatment with immunotherapy (alone or in combination with chemotherapy) for metastatic disease by investigators' choice within the framework of good clinical practice and in agreement with current guidelines;
* Will to participate by providing written informed consent;
* Availability to administer oral supplements and immunotherapy with or without chemotherapy;
* Eastern Cooperative Oncology Group Performance Status ≤ 2;
* Life expectancy ≥ 6 months.

Exclusion Criteria:

* Age < 18 years;
* Inability to sign an informed consent;
* Indication to or ongoing artificial nutrition support (totally compromised spontaneous food-intake) and incapacity or unavailability to consume oral nutritional supplements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 12 months
  A progression-free survival rate at 12 months will be calculated, with patients categorized in a dichotomous manner as alive and progression-free or in progression or dead at 12 months.

SECONDARY OUTCOMES:
Duration of response | 24 months
  Time to progression
Overall survival | 24 months
  Overall survival
Treatment-related moderate-severe adverse events as assessed by Common Terminology Criteria for Adverse Events [CTCAE v5.0] | 4 months
  Difference in the incidence of grade >=3 toxicity, according to CTCAE v5.0
Skeletal muscle mass | 12 months
  Change in skeletal muscle mass during the study evaluated with bioimpedance vectorial analysis and computed tomography scans
Fatigue | 12 months
  Change in fatigue during the study as assessed by the Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) questionnaire
Self-perceived quality of life | 12 months
  Change in quality of life during the study as assessed by validated questionnaires
Self-reported physical activity level | 12 months
  Change in self-reported physical activity level as assessed by the Godin's Shepard Leisure Time Exercise Questionnaire

OTHER OUTCOMES:
Serum levels of immunologic markers | 12 months
  Change in levels of soluble effectors and immuno-regulatory cells during the study by cytofluorimetry and validated biochemical assays

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Caccialanza, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Depending on a specific research question and according to a study protocol to be approved by the Ethics Committee

REFERENCES:
- [Derived] Caccialanza R, Cereda E, Agustoni F, Klersy C, Casirati A, Montagna E, Carnio S, Novello S, Milella M, Pilotto S, Trestini I, Buffoni L, Ferrari A, Pedrazzoli P. Multicentre, randomised, open-label, parallel-group, clinical phase II study to evaluate immunonutrition in improving efficacy of immunotherapy in patients with metastatic non-small cell lung cancer, undergoing systematic nutritional counseling. BMC Cancer. 2022 Nov 24;22(1):1212. doi: 10.1186/s12885-022-10296-x. PMID 36434615